CLINICAL TRIAL: NCT06443723
Title: Metabolic Dysfunction Associated Fatty Liver Disease in Long-Term Cholecystectomy: A Cross-sectional Case-control Study
Brief Title: Metabolic Dysfunction Associated Fatty Liver Disease in Long-Term Cholecystectomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Semih Sezer, Principal Investigator, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CholecystectomyMAFLD
Record Dates: First submitted 2024-05-19; First posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Liver Steatoses
Keywords: Ultrasaund; obesity; cholecystectomy
MeSH Terms: conditions — Fatty Liver; Obesity | interventions — Hematologic Tests; Body Height; Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cholecystectomy (Experimental): Evaluation of hepatosteatosis by hepatobiliary ultrasonography in cholecystectomy patients. Height, hip, waist circumference, blood pressure measurement and hemogram, lipid parameters.
  Interventions: Diagnostic Test: USG, blood tests, waist, hip, height and blood pressure measurements
- Control (Experimental): Evaluation of hepatosteatosis by hepatobiliary ultrasonography in participants without cholecystectomy. Height, hip, waist circumference, blood pressure measurement and hemogram, lipid parameters.
  Interventions: Diagnostic Test: USG, blood tests, waist, hip, height and blood pressure measurements

INTERVENTIONS:
Diagnostic Test: USG, blood tests, waist, hip, height and blood pressure measurements — MAFLD is defined as hepatic steatosis entity in addition to the presence of overweight or obesity, DM, or evidence of metabolic dysfunction.
  Metabolic dysfunction (two or more of the following)
  1. waist circumference ≥ 90 cm in men and 88 cm in women,
  2. blood pressure ≥ 130/85 mmHg or on specific drug treatment,
  3. plasma triglycerides (TG) ≥ 150 mg/dl or on specific drug treatment,
  4. plasma high-density lipoprotein cholesterol (HDL-C) < 40 mg/dl for men and 50 mg/dl for women or on specific drug treatment,
  5. prediabetes (FBS 100 to 125 mg/dl or HbA1c 5.7 to 6.4%),
  6. homeostasis model assessment of insulin resistance (HOMA-IR) score ≥ 2.5.

SUMMARY:
The aim of this study was to examine the association between metabolic associated fatty liver disease (MAFLD) in participants who had undergone cholecystectomy and those who had not undergone cholecystectomy. MAFLD is defined as hepatic steatosis(with ultrasonography) entity in addition to the presence of overweight or obesity, diabetes mellitus, or evidence of metabolic dysfunction.

In this way, the long-term effects of cholecystectomy surgeries, which are commonly performed in the society and thought to be harmless, will be evaluated.

DETAILED DESCRIPTION:
Cholecystectomy is known to be a harmless operation with low perioperative mortality and morbidity. However, the unexplained increase in metabolic disorders in cholecystectomy patients has led to the need for further investigation of cholecystectomy patients. Non-alcoholic fatty liver disease is an important health problem with an average prevalence of 25% worldwide and serious hepatic and systemic complications. The aim of this study was to examine the association of cholecystectomy with metabolic dysfunction associated fatty liver disease (MAFLD), which is an important public health problem in the long-term.

This case-controlled cross-sectional study was planned to evaluate the relationship between patients who had undergone cholecystectomy with MAFLD. MAFLD is defined as hepatic steatosis entity in addition to the presence of overweight or obesity, diabetes mellitus, or evidence of metabolic dysfunction.

The study included 86 participants with cholecystectomy and 63 participants without cholecystectomy. It was planned to compare the participants according to the diagnostic criteria for MAFLD (with or without MAFLD).

ELIGIBILITY:
Inclusion Criteria:

* who were found to have undergone cholecystectomy at least five years ago,
* who could feed orally and perform activities of daily living
* participants who had not undergone cholecystectomy with similar characteristics were included in the study

Exclusion Criteria:

* those with chronic liver disease
* malignancy or history of malignancy
* in a chemotherapy program
* with active infection
* any organ failure
* pregnancy
* use of drugs that cause steatosis in the liver

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
diabetes mellitus | through study completion, an average of 4 months
  fasting plasma glucose >126mg/dL
definition of overweight | through study completion, an average of 4 months
  BMI >25 kg/m2
Upper limits of waist circumference | through study completion, an average of 4 months
  ≥102 cm in men and 88 cm in women
Definition of pre-diabetes | through study completion, an average of 4 months
  fasting plasma glucose of 100-125 mg/dL
Blood pressure upper limit | through study completion, an average of 4 months
  ≥130/85 mmHg
HDL-cholesterol levels | through study completion, an average of 4 months
  <40 mg/dL for males and <50 mg/dL for females.
Triglyceride levels | through study completion, an average of 4 months
  ≥1.70 mmol/L
Diagnosis of MAFLD | through study completion, an average of 4 months
  hepatic steatosis + (diabetes mellitus and/or overweight and/or metabolic dysfunction) metabolic dysfunction is defined as the presence of at least two criteria(Pre-diabetes, TG, HDL, blood pressure, waist circumference)

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)